CLINICAL TRIAL: NCT04080102
Title: Metabolic Effects of Essential Amino Acids and High-intensity Interval Training
Brief Title: Essential Amino Acids and High Intensity Interval Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Strength and Conditioning Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-2726
Record Dates: First submitted 2019-08-26; First posted 2019-09-06 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Risk Factor; Obesity
MeSH Terms: conditions — Obesity | interventions — High-Intensity Interval Training; Amino Acids, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High intensity interval training (HIIT) (Experimental)
  Interventions: Other: High Intensity Interval Training
- Essential Amino Acid Supplement (Experimental)
  Interventions: Dietary Supplement: Essential Amino Acid
- High intensity interval training + Essential Amino Acid (Experimental)
  Interventions: Other: High intensity interval training and essential amino acid supplement
- Control (No Intervention)

INTERVENTIONS:
Other: High Intensity Interval Training — Exercise
  Arms: High intensity interval training (HIIT)
Dietary Supplement: Essential Amino Acid — Oral ingestion of a powdered dietary supplement
  Arms: Essential Amino Acid Supplement
Other: High intensity interval training and essential amino acid supplement — Exercise and dietary supplement
  Arms: High intensity interval training + Essential Amino Acid

SUMMARY:
Purpose: The primary purpose is to determine the combined effects of essential amino acids (EAA) supplementation and high intensity interval training (HIIT) on body composition, muscle characteristics, and muscle architecture in overweight men and women over the course of eight weeks. A secondary purpose is to determine the metabolic effects of EAA supplementation and HIIT on whole body protein turnover, metabolic rate, substrate metabolism, and metabolomics. A tertiary purpose is to evaluate the modulatory effects of sex on body composition, metabolism, metabolic profile, cardiorespiratory fitness, and hunger and satiety in response to EAA supplementation and HIIT. Participants: Healthy overweight and obese men and women (30-50 years) Procedures (methods): In a block randomized design, 78 healthy, overweight or obese men and women will be randomized, to one of four, eight-week intervention groups using a 2:2:2:1 group allocation design: 1) essential amino acids (EAA) supplementation (7.2 grams EAA daily); 2) HIIT, two days per week of cycle ergometry training; 3) EAA + HIIT; or 4) control (CON), receiving no intervention. Measurements of body composition, muscle characteristics, resting metabolic rate, substrate metabolism, and cardiorespiratory fitness will be measured at baseline, 4-weeks, and 8-weeks. Metabolomics and whole body protein turnover will also be measured at baseline and 8-weeks. Subjects will be asked to arrive to testing sessions following a 12 hour fast (except for water), consuming no food, caffeine, or alcohol. Participants will also be asked to abstain from physical activity for 24 hours prior to testing. Subjects will complete one electronic contact (phone/email screening) and up to 22 in-person sessions (enrollment; 5 testing sessions [2 at base, 1 at 4week, 2 at 8week]; 16 training sessions [for HIIT and EAA+HIIT]) over the course of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (25-50 years).
* Overweight and obese: body mass index (BMI) of 27 - 40 kg·m-2 and/or percent body fat > 25% for men, and BMI of 25 - 40 kg·m-2 and/or Percent Body Fat > 30% for women.
* Healthy, non-smokers.
* Women: eumenorrheic, reporting consistent menstruation, having 3 regular cycles in the 3 months prior to enrollment, and not pregnant or planning on becoming pregnant.

Exclusion Criteria:

* Have current and/or history of cardiovascular disease, diabetes, metabolic, thyroid, pulmonary, renal, hepatic, gastrointestinal, musculoskeletal disorders or medical or surgical events, such as bariatric surgery, heart surgery, or any joint or musculoskeletal surgeries occurring in the 6-months prior to enrollment, that may significantly influence study outcomes or prevent safe participation.
* Have uncontrolled hypertension or an abnormal electrocardiogram.
* Have a diagnosed mental disorder
* Inconsistently taking medications or taking medications that may influence study outcomes.
* Participating in more than 150 minutes per week of moderate exercise, more than 2 days per week of resistance training, or currently participating in high intensity interval training or participated in HIIT within the previous 12 weeks.
* Lost or gained greater than eight pounds within three months prior to the enrollment.
* Currently consuming a high protein diet (,1.6 g·kg-1·day-1 and <25% of calories from protein).
* Currently consuming meal replacements or dietary supplements that may taurine, or beta-hydroxy beta-methylbutyrate) within eight weeks prior to the enrollment date.
* Reports any known sensitivity to the Essential Amino Acid treatment.
* Has participated in another clinical trial within four weeks prior to enrollment that in the opinion of the PI would influence the results.
* Has severely impaired hearing or speech or inability to speak English.
* Unwilling or unable to comply with the study protocol, including abstaining from, caffeine, tobacco, alcohol, and physical activity before testing days.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-01-05 (Actual)

PRIMARY OUTCOMES:
Fat Free Mass (kg) | 8 weeks
  Determined from a multi-compartment model
Fat mass (kg) | 8 weeks
  Determined from a multi-compartment model

SECONDARY OUTCOMES:
Muscle cross sectional area (cm3) | 8 weeks
  Determined from ultrasound
Echo intensity (a.u.) | 8 weeks
  Determined from ultrasound

OTHER OUTCOMES:
Metabolic rate (kcal/day) | 8 weeks
  resting metabolic rate from indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Study Director — University of North Carolina, Chapel Hill; Katie Hirsch, MA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Applied Physiology Laboratory, Fetzer Hall Room 25, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 24 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina (UNC).
Time Frame: Deidentified individual data that supports the results will be shared beginning 12 to 24 months following publication.
Access Criteria: An investigator who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Hirsch KR, Greenwalt CE, Cabre HE, Gould LM, Brewer GJ, Blue MNM, Ferrando AA, Huffman KM, Mayer-Davis EJ, Ryan ED, Smith-Ryan AE. Metabolic effects of high-intensity interval training and essential amino acids. Eur J Appl Physiol. 2021 Dec;121(12):3297-3311. doi: 10.1007/s00421-021-04792-4. Epub 2021 Aug 24. PMID 34427732